CLINICAL TRIAL: NCT04902001
Title: Role of Mechanical Load on Metabolic Exercise Adaptations in Response to Weight Loss in Obese Adolescents: The POWELL Study
Acronym: POWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2021 BOIRIE; 2021-A00756-35 (Other: 2021-A00756-35)
Record Dates: First submitted 2021-05-03; First posted 2021-05-26 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Pediatric Obesity
Keywords: energy expenditure; weight loss; obesity; adolescents
MeSH Terms: conditions — Pediatric Obesity; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: One group of adolescents with obesity
Masking Description: There is no need for masking here.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with obesity (Experimental): Adolescents with obesity aged 12-16 years old
  Interventions: Behavioral: Multidisciplinary weight loss

INTERVENTIONS:
Behavioral: Multidisciplinary weight loss — The adolescents will follow a 12-week intervention combining nutritional education, physical activity 3 times per week and psychological supports.

SUMMARY:
While interdisciplinary weight loss intervention have been shown successful among adolescents with obesity, a weight regain is most of the time observed within the following weeks or months. The aim of the present project will be to better identify the independent role played by both the metabolic and mechanical load and their modification during weight loss, on the energy expenditure and energy metabolism of adolescents with obesity.

DETAILED DESCRIPTION:
A total of 28 adolescents with obesity will be recruited from our local inpatient pediatric obesity centers. Before their weight loss intervention the adolescents will complete two experimental visits. During the first visit, anthropometric and body composition measurements will be performed. Then the participants will be asked to complete a walking exercise on a treadmill during the second visit. Their energy expenditure and substrate oxidation will be assessed by indirect calorimetry. They will have to walk at 5 different walking speeds. Then, they will follow a 12-week weight loss intervention. By the end of this intervention, their body composition will be assessed and they will be asked to perform the same walking exercise. On a separate occasion (randomly assigned) they will have to repeat this walking exercise while carrying a load corresponding of their weight loss.

ELIGIBILITY:
Inclusion Criteria:

* being aged 12-16 years old
* no contraindication to physical exercise
* no cardiovascular disease
* BMI above the 97th percentile
* candidate to a weight loss intervention

Exclusion Criteria:

* surgery and medical conditions preventing them to perform the intervention
* Weight loss during the previous 6 months
* medication that could interfere with energy metabolism.
* pregnancy
* regular tobacco and alcool use

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Change in Energy Expenditure between before and after weight loss | before and after the 12-week weight loss
  amount of energy expended during the walking tests, measured using indirect calorimetry

SECONDARY OUTCOMES:
change in lipid oxidation between before and after weight loss | before and after the 12-week weight loss
  amount of lipids oxidized during the walking tests, measured using indirect calorimetry
change in Fat mass between before and after weight loss | before and after the 12-week weight loss
  The amount of body fat will be assessed by dual energy X-ray absorptiometry
change physical activity preferences between before and after weight loss | before and after the 12-week weight loss intervention
  Children will be asked to indicate their prefered physical activties and sedenatry behaviors on a computer task using visual analog scale (from 0 to 150 mm)
Change in Energy Expenditure between the unloaded and loaded walking test | after the 12_week weight loss
  amount of energy expended during the walking tests, measured using indirect calorimetry
Change in lipid oxidation between the unloaded and loaded walking test | after the 12_week weight loss
  amount of lipids oxidized during the walking tests, measured using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France